CLINICAL TRIAL: NCT05487261
Title: Pulmonary REsistance Modification Under Treatment With Sacubitril/valsartaN in paTients With Heart Failure With Reduced Ejection Fraction - PRESENT HF Study
Brief Title: Pulmonary REsistance Modification Under Treatment With Sacubitril/valsartaN in paTients With Heart Failure With Reduced Ejection Fraction
Acronym: PRESENT-HF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Hospital Heliodor Swiecicki of the Medical University of Karol Marcinkowski in Poznań (Other)
Collaborators: Medical Research Agency, Poland (Other Government); Medical University of Bialystok (Other); University of Opole (Other); Medical University of Gdansk (Other); Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/ABM/01/00078
Record Dates: First submitted 2022-07-26; First posted 2022-08-04 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril and valsartan combination (Experimental): Patient receive: 1 bottle with Sacubitril/Valsartan tablets and 2nd bottle with placebo to enalapril.
  Interventions: Drug: Sacubitril-valsartan; Drug: Placebo
- Enalapril (Active Comparator): Patient receive: 1 bottle with placebo to Sacubitril/Valsartan and 2nd bottle with enalapril.
  Interventions: Drug: Enalapril; Drug: placebo

INTERVENTIONS:
Drug: Sacubitril-valsartan — level 1-24 / 26mg 2 times a day, level 2-49 / 51mg 2 times a day, level 3-97 / 103mg 2 times aday
  Arms: Sacubitril and valsartan combination
Drug: Enalapril — level 1-2.5 mg twice a day, level 2-5 mg twice a day, level 3-10 mg twice a day
  Arms: Enalapril
Drug: placebo — placebo matching for 24 / 26mg, 49 / 51mg, 97 / 103mg 2 of sacubitril/valsartan
  Arms: Enalapril
Drug: Placebo — placebo matching for 2.5 mg, 5 mg, 10 mg of enalapril
  Arms: Sacubitril and valsartan combination

SUMMARY:
MAIN OBJECTIVE. Demonstration that use of sacubitril/valsartan influences parameters of right heart catheterization, including pulmonary artery pressure, and provokes changes in pulmonary circulation resistance in patients with heart failure with reduced left ventricular ejection fraction (HFrEF) and post-capillary pulmonary hypertension (PH): both isolated post-capillary (Ipc-PH) and combined post- and pre-capillary (Cpc-PH), which we predict could improve prognosis in this group of patients.

RESEARCH HYPOTHESIS. Sacubitril/valsartan used in patients with HFrEF accompanied by pulmonary hypertension due to HFrEF will reduce pulmonary artery pressure, pulmonary vascular resistance, and the incidence of secondary end-points as listed in the protocol.

STUDY OUTLINE. PRESENT-HF will show the effects of sacubitril/valsartan on pulmonary circulation pressure in patients with HFrEF and post-capillary pulmonary hypertension (PH): both isolated post-capillary (Ipc-PH) and combined post- and pre-capillary (Cpc-PH), which is expected to improve prognosis.

DETAILED DESCRIPTION:
Non commercial, multicentre, randomised, double-blind, comparator-controlled clinical trial. Eligible patients were randomly assigned (1:1) using a secure, central, interactive, web-based response system, to intervention or comparator arm. Time of observation 13 months [1months active up titration phase + 12 months follow up].

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age who are able to complete and sign the informed consent form.
2. HF patients in NYHA functional class II-IV with a reduced left ventricular ejection fraction (LVEF) ≤40% -(HFrEF) (confirmed by an examination such as echocardiography or cardiac magnetic resonance within the last 6 months) in whom right heart catheterization (RHC) reveals post-capillary or mixed pulmonary hypertension (defined on the basis of the 2015 ESC (European Society of Cardiology) guidelines: mean pulmonary artery pressure (PAPm) ≥25 mmHg and pulmonary capillary wedge pressure (PCWP)>15mmHg) were found, both of the isolated extracapillary PH (Ipc-PH) (defined on the basis of the 2015 ESC guidelines: DPG < 7 mm Hg and / or PVR ≤ 3 WU) as well as complex extra-and pre-capillary PH (Cpc-PH) (defined on the basis of the 2015 ESC guidelines: DPG ≥ 7 mm Hg and / or PVR> 3 WU).
3. Stable patients haemodynamics, which is defined as no change in diuretic use for at least 4 weeks prior to study entry.
4. HF during optimal treatment with ACE-I (angiotensin converting enzyme) /ARB (angiotensin receptor blocker), beta blocker, MRA (Mineralocorticoid Receptor Antagonists), SGLT2-I except in cases where the above-mentioned treatment was contraindicated or not tolerated.
5. Understanding and acceptance of the research assumptions and methods and signing the informed consent by the patient.

Exclusion Criteria:

1. Current treatment with S/V.
2. Cardiogenic shock.
3. Current treatment with sildenafil.
4. Patients ineligible or contraindicated for treatment with sacubitril-valsartan.
5. Patients with a history of angioedema.
6. Patients who have had a heart transplant or have had a circulatory support device.
7. Patient on the urgent list for heart transplant.
8. Isolated right HF secondary to lung disease.
9. Documented untreated significant ventricular arrhythmia with syncope within the previous 3 months.
10. Symptomatic bradycardia or second or third degree atrioventricular block not protected by a pacemaker.
11. Factors that prevent RHC testing (e.g. very serious condition of the patient that makes it impossible to lie down, cardiogenic shock, allergy to contrast agents, etc.).
12. Pregnant or lactating women.
13. Women of childbearing age, defined as the physiological possibility of becoming pregnant, unless using two methods of contraception.
14. Acute coronary syndrome, including myocardial infarction (STEMI, NSTEMI), a condition with carotid revascularization or major cardiovascular surgery in the last 30 days.
15. Stroke or transient cerebral ischemia (TIA) within the last 3 months.
16. Previous CRT (Cardiac Resynchronization Therapy) implantation in the last 3 months or planning for CRT implantation.
17. Life expectancy <6 months.
18. Severe renal failure, eGFR (epidermal growth factor receptor) <30 ml / min / 1.73 m2(calculated according to the MDRD formula).
19. Serum potassium> 5.2 mEq/L.
20. Liver failure or elevated liver transaminases (total bilirubin> 3 mg / dL and/or ALT (Aspartate transaminase) and/or AST (Aspartate Aminotransferase) ≥3x ULN).
21. A major surgery planned within 6 months of randomization.
22. Planned coronary angioplasty or pacemaker / ICD (implantable cardioverter defibrillator) / CRT implantation within the next 6 months.
23. Severe primary valve disease (NOT secondary mitral regurgitation) or obstructive hypertrophic cardiomyopathy.
24. The presence of a malignant neoplasm of any organ system, ie clinical signs or no stable remission for at least 3 years after the end of the last treatment, with the exception of non-invasive basal cell carcinoma, squamous cell carcinoma of the skin or cervical epithelial dysplasia.
25. Diseases that significantly reduce physical performance:

    1. severe COPD (chronic obstructive pulmonary disease) putting off oxygen therapy,
    2. severe asthma,
    3. morbid obesity (BMI> 40 kg / m2),
    4. significant lower limb atherosclerosis with intense intermittent claudication.
26. Uncontrolled hypertension (SBP> 170 mmHg and / or DBP> 100 mmHg).
27. Symptomatic hypotension (SPB <90 mmHg)
28. Any situation that may make it impossible to perform the research in accordance with the protocol or express written consent in the opinion of the researcher, including abuse of alcohol, drugs or other psychoactive substances.
29. Participation in a study with a device or medicinal product within 3 months prior to randomization or 5 half-lives, whichever is longer, prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
mean pulmonary artery pressure | 0-13 month
  change from baseline in mean pulmonary artery pressure (mPAP), measured invasively in Right Heart Catheterization (RHC)
pulmonary vascular resistance | 0-13 month
  change from baseline in pulmonary vascular resistance (PVR), calculated from data measured invasively in Right Heart Catheterization (RHC)

SECONDARY OUTCOMES:
pulmonary wedge pressure | 0 -13 month
  change from baseline in pulmonary wedge pressure (PWP), measured invasively in Right Heart Catheterization (RHC)
diastolic pressure gradient | 0-13 month
  change from baseline in the diastolic pressure gradient (DPG; where DPG = diastolic mPAP -mean PWP)
6-minute walk test | 0-13 month
  change in the 6-minute walk test (6MWT) - analysis of changes from the baseline
spiroergometric test (CPET, Cardio-Pulmonary Exercise Test) | 0-13 month
  evaluation of the parameters of the spiroergometric test - analysis of changes in relation to the baseline
echocardiographic parameters | 0-13 month
  assessment of echocardiographic parameters - analysis of changes in echocardiographic parameters assessed in transthoracic echocardiographic examination (TTE)
composite endpoint of MACCEs (major adverse cardiac and cerebrovascular events) | 0-13 month
  The incidence of the composite endpoint of MACCEs such as death from all causes, cardiac death, hospitalization due to worsening/ decompensation of heart failure (HF), stroke/ transient ischemic attack (TIA), acute coronary syndrome (ACS), the need for a heart transplant (HT), the need for a left ventricular assist device (LVAD) or biventricular(BVAD)
hospitalization or an unplanned visit to the Emergency Department | 0-13 month
  hospitalization or an unplanned visit to the Emergency Department or an unplanned outpatient visit related to HF
unplanned intravenous administration of diuretics and/or an unplanned hospitalization | 0-13 month
  the need for unplanned intravenous administration of diuretics and/or an unplanned hospitalization, outpatient visit due to the need to administer intravenous diuretics or requiring an increase in the dose of diuretics >50% from baseline
quality of life measurements - Short Form 36 Health Survey (SF-36 questionnaire) | 0-13 month
  assessment of quality of life - SF-36 questionnaire - change from the baseline, the minimum and maximum values: 0-100, higher scores mean a less disability.
quality of life measurements - Kansas City Cardiomyopathy Questionnaire (KCCQ) | 0-13 month
  assessment of quality of life - KCCQ, the minimum and maximum values: 0-100, higher scores mean higher quality of life.
quality of life measurements - EuroQol-5 Dimensions-3 Level (EQ-5D-3L) questionnaire | 0-13 month
  assessment of quality of life - EQ-5D-3L questionnaire - change from the baseline, the minimum and maximum values: 0-100, higher scores mean higher quality of life.
quality of life measurements - The World Health Organization Quality of Life (WHOQOL) | 0-13 month
  assessment of quality of life - WHOQOL - change from the baseline, the minimum and maximum values: 0-100, higher scores mean higher quality of life.
the New York Heart Association functional classes | 0-13 month
  assessment of the New York Heart Association (NYHA) functional classes - change from the baseline, the minimum and maximum values: 1-4, higher scores mean a worse outcome.
the World Health Organization functional classes | 0-13 month
  assessment of the World Health Organization (WHO) functional classes - change from the baseline, the minimum and maximum values: 1-4, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Straburzyńska-Migaj, Prof. MD, Principal Investigator — University Hospital in Poznan
Locations (5):
- Poland (5):
  - Medical University of Bialystok Clinical Hospital, Bialystok
  - University Clinical Centre in Gdańsk, Gdansk
  - University Clinical Hospital in Opole, Opole
  - University Hospital in Poznan, Poznan
  - Specialist Hospital in Zabrze, Zabrze